CLINICAL TRIAL: NCT04361136
Title: A Phase 1 Clinical Trial to Evaluate the Phototoxic Potential of Delgocitinib Cream After Single Topical Occlusive Application on Healthy Skin
Brief Title: Clinical Trial to Evaluate Light-induced Skin Reactions After Application of Delgocitinib Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LP0133-1408; 2019-000705-67 (EudraCT Number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: All subjects will receive all treatments with treatments randomised over test fields.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Delgocitinib cream 1 mg/g (Experimental): Single topical occlusive administration
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 3 mg/g (Experimental): Single topical occlusive administration
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 8 mg/g (Experimental): Single topical occlusive administration
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 20 mg/g (Experimental): Single topical occlusive administration
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream vehicle (Placebo Comparator): Single topical occlusive administration
  Interventions: Drug: Delgocitinib cream vehicle

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application
  Other Names: LEO 124249 cream
  Arms: Delgocitinib cream 1 mg/g; Delgocitinib cream 20 mg/g; Delgocitinib cream 3 mg/g; Delgocitinib cream 8 mg/g
Drug: Delgocitinib cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
  Other Names: LEO 124249 cream vehicle
  Arms: Delgocitinib cream vehicle

SUMMARY:
This is a single-centre, randomised, vehicle-controlled, double-blind, within-subject comparison phase 1 clinical trial. The trial is designed to find out if delgocitinib cream can cause skin irritation after light exposure in people with healthy skin.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy subjects aged 18-64 years (inclusive).
* Fitzpatrick skin type of I, II, or III.

Key Exclusion Criteria:

* Atopic dermatitis, eczema, psoriasis, acne, dermatitis solaris or suntan that could interfere with the test field evaluation, hyperpigmentation, multiple naevi, tattoos, blemishes or dense body hair in the range of the test fields.
* Any history of or presence of cancerous or precancerous skin lesions.
* Any other skin disease or other visible skin condition noted on physical examination which in the investigator's opinion might interfere with the evaluation of the test field reaction.
* Known disease that can be induced by ultraviolet (UV) light.
* Use of any topical or systemic medication which could interfere with the trial objective within 2 weeks before randomisation until end of trial.
* Use of drugs which might cause photobiologic or phototoxic reactions within 4 weeks before randomisation until end of trial.
* Foreseeable intensive UV light exposure (solar or artificial) to test fields within 4 weeks before randomisation until end of trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Positive skin reaction at 24 hours or 48 hours after irradiation | Up to 48 hours after irradiation
  A reaction is considered positive if the skin reaction score for the irradiated test field is at least 1 point higher than both the non-irradiated test field exposed to the same strength of IMP, and the irradiated control field.
  The grading for the skin reaction score will be performed according to the following 5-point scale:
  * 0 No reaction
  * 1 Erythema
  * 2 Erythema with dermal infiltrate
  * 3 Erythema with papulovesicles
  * 4 Erythema with blisters, erosions

SECONDARY OUTCOMES:
Positive skin reaction at 24 hours after irradiation | 24 hours after irradiation
  A reaction is considered positive if the skin reaction score for the irradiated test field is at least 1 point higher than both the non-irradiated test field exposed to the same strength of IMP, and the irradiated control field.
  The grading for the skin reaction score will be performed according to the following 5-point scale:
  * 0 No reaction
  * 1 Erythema
  * 2 Erythema with dermal infiltrate
  * 3 Erythema with papulovesicles
  * 4 Erythema with blisters, erosions
Positive skin reaction at 48 hours after irradiation | 48 hours after irradiation
  A reaction is considered positive if the skin reaction score for the irradiated test field is at least 1 point higher than both the non-irradiated test field exposed to the same strength of IMP, and the irradiated control field.
  The grading for the skin reaction score will be performed according to the following 5-point scale:
  * 0 No reaction
  * 1 Erythema
  * 2 Erythema with dermal infiltrate
  * 3 Erythema with papulovesicles
  * 4 Erythema with blisters, erosions

OTHER OUTCOMES:
Number of treatment-emergent adverse events from baseline to Day 4 | From time of first investigational medicinal product application (Day 1) until Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Bioskin Research Center Dermatology, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No